CLINICAL TRIAL: NCT05122429
Title: Asynchronous Techniques for the Delivery of Empirically Supported Psychotherapies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Adam Gonzalez, Associate Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NNX15AN64G
Record Dates: First submitted 2021-10-18; First posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Depressive Symptoms; Anxiety; Stress; Impairment
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- myCompass Only (Experimental): Self-guided e-health treatment
  Interventions: Behavioral: e-Health Treatment
- myCompass + Delayed Text Therapy Support (Experimental): Self-guided e-health treatment with delayed (44min) text support from a therapist.
  Interventions: Behavioral: e-Health Treatment
- myCompass + Delayed Video Therapy Support (Experimental): Self-guided e-health treatment with delayed (44min) video support from a therapist.
  Interventions: Behavioral: e-Health Treatment

INTERVENTIONS:
Behavioral: e-Health Treatment — Self-guided e-health treatment with two of the arms providing delayed (44min) text or video support from a therapist.

SUMMARY:
The aim of this study is to test the feasibility, acceptability and efficacy of methods for delivering mental health support when real-time communication is not possible (e.g. on long duration space flights where communication lags of up to 45 minutes are anticipated). The investigators hypothesize that the two enhanced treatment conditions (i.e., those with therapist support) will outperform the online self-management program without support. The investigators also predict that outcomes for the two enhanced conditions will be comparable to those reported in the literature for in-person psychotherapy programs.

DETAILED DESCRIPTION:
The aim of this study is to test the feasibility, acceptability and efficacy of methods for delivering mental health support when real-time communication is not possible (e.g. on long duration space flights where communication lags of up to 45 minutes are anticipated). Participants will be healthy, high functioning adults (e.g., medical residents, postdoctoral fellows in the sciences, math, and engineering) who report elevated psychological distress, mood or anxiety symptoms. Participants will complete a self-guided online therapy program (MyCompass) and will be randomized to receive one of the following: (1) online therapy without therapist support, 2) online therapy plus therapist support via electronic text-based messaging (i.e., secure email), or 3) online therapy plus therapist support via video messaging. Outcomes will be evaluated weekly via online self-report measures of psychological distress, mood, anxiety, number of hours and quality of sleep, fatigue, and resiliency indicators (i.e., coping and mindfulness). The investigators will examine changes over time in outcomes across all three groups. The investigators hypothesize that the two enhanced treatment conditions (i.e., those with therapist support) will outperform the online self-management program without support. The investigators also predict that outcomes for the two enhanced conditions will be comparable to those reported in the literature for in-person psychotherapy programs.

ELIGIBILITY:
Inclusion Criteria:

1. 18+years old;
2. Masters of Art degree or higher in social/biomedical(medicine)/physical science, engineering or mathematics
3. current elevated distress as measured by the Depression Anxiety and Stress Scale, 21 item version(≥ 5 on DASS Depression Subscale OR ≥ 4 on DASS Anxiety Subscale OR ≥ 8 on DASS Stress Subscale) (DASS, Lovibond & Lovibond, 1995); and, (5) ≥ 5 on any subscale of the Sheehan Disability Scale (SDS, Sheehan 1983).

Exclusion Criteria:

1. Any current or recent (i.e. past month) suicide ideation
2. any history of suicide attempt (within past 5 years)
3. serious mental illness (i.e., psychosis, mania)
4. alcohol or substance dependency during the past 6 months
5. serious medical problems (e.g., seizures, cancer)
6. current participation in psychotherapy
7. new use of psychoactive medications (i.e., benzodiazepines for less than 1 month or selective serotonin reuptake inhibitors [SSRIs], tricyclics, or serotonin-norepinephrine reuptake inhibitors [SNRIs] for less than 3 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Functional impairment in work/school, social life, and family life change | Change from baseline at 6-weeks assessments, 1-weeks post treatment, and 1-month post treatment
  Sheehan Disability Scale is a 3 item measure to assess functional impairment in work/school, social life, and family life.
Symptoms of Depression, Stress, and Anxiety Change | Change from baseline at 6-weeks assessments, 1-week post treatment, and 1-month post treatment
  Depression Anxiety and Stress Scale is a 21-item measure to assess the severity of Depression, Stress, and Anxiety.

SECONDARY OUTCOMES:
Sleep Quality Change | Change from baseline at 1-week post treatment and 1-month post treatment
  The Pittsburgh Sleep Quality Index (PSQI) is a 19-item questionnaire that assesses seven components of sleep quality (subjective sleep quality, sleep latency, duration, efficiency, disturbances, use of sleep medication, and daytime dysfunction). Each component is rated on a 0-3 severity scale referring to the frequency of each disturbance, and yields a global score with a range of 0-21.
Fatigue Severity Change | Change from baseline at 1-week post treatment and 1-month post treatment
  The Fatigue Severity Scale (FSS) measures fatigue and its effects on functioning. The FSS is comprised of nine items rated on a Likert-type rating scale (1-7), where one indicates no impairment and seven indicates severe impairment.
Treatment Satisfaction | 1-week post treatment
  The ARMS-12 measures confidence, comfortability, and perceptions towards the program. The ARMS-12 is comprised of 12 items rated on a Likert-type rating scale (1-7), where one indicates the how strongly the agree or disagree with the statement.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Gonzalez, PHD, Principal Investigator — Stony Brook University
Locations (1):
- Mind-Body Clinical Research Center, Stony Brook, New York, United States

REFERENCES:
- [Derived] Luo X, Bugatti M, Molina L, Tilley JL, Mahaffey B, Gonzalez A. Conceptual Invariance, Trajectories, and Outcome Associations of Working Alliance in Unguided and Guided Internet-Based Psychological Interventions: Secondary Analysis of a Randomized Controlled Trial. JMIR Ment Health. 2022 Jun 21;9(6):e35496. doi: 10.2196/35496. PMID 35727626